CLINICAL TRIAL: NCT05902390
Title: A Prospective, Multicenter, Exploratory Clinical Study to Evaluate the Long-term Benefit of Hydrogel Spacer in Reducing Rectal Radiation Dose in Cervical Cancer Radiation Therapy.
Brief Title: The Long-term Benefit of Hydrogel Spacer in Reducing Rectal Radiation Dose in Cervical Cancer Radiation Therapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Shanghai Reunion Biotech Co.,Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RN-CT-003
Record Dates: First submitted 2023-06-05; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Cervical Cancer; hydrogel spacer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hydrogel spacer (Experimental): The Subjects randomized to the treatment group underwent placement of hydrogel spacer.
  Interventions: Device: hydrogel spacer
- Control (No Intervention): The Subjects randomized to the control group did not receive injection of the hydrogel spacer.

INTERVENTIONS:
Device: hydrogel spacer — Randomly assigned to either the treatment group, who were injected with hydrogel spacer, or the control group, who were not injected with hydrogel spacer.
  Arms: hydrogel spacer

SUMMARY:
This study is an exploratory study based on the previous study " A prospective, multicenter, randomized, parallel arm-controlled, superiority clinical study to evaluate the role of hydrogel spacer in reducing rectal radiation dose in cervical cancer radiation therapy", in which additional follow up study on the subjects of the previous study were conducted. Subjects (6 subjects in Phase I; 100 subjects in Phase II, 50 in the test group and 50 in the control group) who completed the pre-study will be enrolled in this study if they are willing to participate in the long-term follow-up by signing the informed consent form.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the long-term benefit of hydrogel spacer when hydrogel is injected between the rectum and cervix in women undergoing radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky score ≥ 70. Subjects aged ≥ 18 years and ≤ 75 years. Subjects must be able to cooperate in completing the entire study. The subjects' pelvic and abdominal cavity and joints are free of metal implants and can tolerate MRI.

No contraindications to CT scanning. Subjects must be able to understand the purpose of the trial, voluntarily participate and sign an informed consent form

Exclusion Criteria:

* Subjects whose target tumors have been previously treated (chemotherapy, immunotherapy, surgical treatment, etc.) Subjects with other primary malignancies Subjects with contraindications to radiotherapy, as determined by the investigators Subjects with injection site infections. Subjects who are allergic to the ingredients of the device. Subjects whose tumors invade the injection site and affect the injection process and injection safety, as determined by the investigators Persons with severe mental illness, cognitive impairment and thinking disorders.

Participants in other drug clinical trials or medical device clinical trials 1 month prior to screening Pregnant or lactating women or those who plan to get pregnant within the last six months Subjects who cannot be followed up as prescribed by the doctor Other conditions that, in the judgment of the investigator, make the subject unsuitable for enrollmen

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
The stability of the hydrogel spacer | Through study completion, an average of 12 months
  In order to verify the stability of the hydrogel spacer, this test will be based on MRI T2-weighed images.
Scores from Quality of Life Questionnaire-Core 30 Rating (QLQ-C30) | through study completion, an average of 12 months
  European Organization for Research on Treatment of Cancer (EORTC) QLQ-C30 is a comprehensive survey instrument designed to assesses the disease-specific aspects of cervical cancer and its therapies. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
Scores from Quality of Life Core Questionnaire Cervix Cancer Module 24 (QLQ-CX24) | through study completion, an average of 12 months
  European Organization for Research on Treatment of Cancer (EORTC) QLQ-CX24 will be used to assess subjects' quality of life. EORTC QLQ-CX24 score from 0 to 100, higher scores indicate better quality of life or more symptoms.
Percentage of subjects with ≥2 grade chronic radiation rectal injury | through study completion, an average of 12 months
  The percentage of subjects in the treatment and control groups who had ≥ grade 2 chronic radiation rectal injury after radiation therapy will be calculated and compared between the groups.
Adverse events requiring special attention | through study completion, an average of 12 months
  The number of cases of adverse events requiring special attention related to radiation intestinal injury and the number of subjects having the above adverse events will be recorded in both the treatment and control groups.
The number of (serious) adverse events, (serious) device-related adverse events | through study completion, an average of 12 months
  The frequency (number of events) of occurrence of (serious) adverse events and device-related (serious) adverse events will be recorded for the entire study period.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] de Freitas AC, Gurgel AP, Chagas BS, Coimbra EC, do Amaral CM. Susceptibility to cervical cancer: an overview. Gynecol Oncol. 2012 Aug;126(2):304-11. doi: 10.1016/j.ygyno.2012.03.047. Epub 2012 Apr 4. PMID 22484226
- [Background] Peach MS, Moore J, Giles W, Trainor J, Long T, Moon N, Hylton JE, Showalter TN, Libby B. Development and preclinical testing of a novel biodegradable hydrogel vaginal packing technology for gynecologic high-dose-rate brachytherapy. J Contemp Brachytherapy. 2018 Aug;10(4):306-314. doi: 10.5114/jcb.2018.77952. Epub 2018 Aug 31. PMID 30237814
- [Background] Kashihara T, Murakami N, Tselis N, Kobayashi K, Tsuchida K, Shima S, Masui K, Yoshida K, Takahashi K, Inaba K, Umezawa R, Igaki H, Ito Y, Kato T, Uno T, Itami J. Hyaluronate gel injection for rectum dose reduction in gynecologic high-dose-rate brachytherapy: initial Japanese experience. J Radiat Res. 2019 Jul 1;60(4):501-508. doi: 10.1093/jrr/rrz016. PMID 31034570